CLINICAL TRIAL: NCT07050992
Title: Laser Posterior Nasal Nerve Neurolysis: a Randonmized Controlled Trial
Brief Title: Laser Posterior Nasal Nerve Neurolysis
Acronym: LPN3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2024071
Record Dates: First submitted 2024-10-10; First posted 2025-07-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Allergic Rhinitis; Chronic Rhinitis; Rhinorrhea; Sneezing; Nasal Obstruction; Nasal Congestion; Nasal Allergies; Nasal Stuffiness
Keywords: laser; posterior nasal nerve; rhinitis; allergy
MeSH Terms: conditions — Rhinitis, Allergic; Rhinorrhea; Sneezing; Nasal Obstruction; Rhinitis; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laser surgery (Active Comparator): Posterior nasal nerve ablation using laser to deliver laser energy to the posterior nasal nerve area.
  Interventions: Procedure: Laser posterior nasal nerve neurolysis
- Sham surgery (Sham Comparator): Sham surgery is performed with the same laser surgical instrument used to enter the nasal cavity for a sham procedure with minimal dosage.
  Interventions: Procedure: Sham surgery

INTERVENTIONS:
Procedure: Laser posterior nasal nerve neurolysis — Posterior nasal nerve ablation using laser is performed through an angled nasal probe at 20 degrees and a 90-degree endoscope to deliver laser energy to the posterior nasal nerve area. The thermal energy is conducted to the middle meatus and the posterior superior part of the inferior turbinate, targeting the area supplied by the posterior nasal nerve. The ablation continues until there is widespread mucosal blanching and the formation of at least one continuous brown eschar
  Arms: Laser surgery
Procedure: Sham surgery — The same laser surgical instrument is used to enter the nasal cavity for a sham procedure with minimal dosage. The energy setting uses the lowest limit of 0.5W with intermittent emission (0.01 second emission with 1 second rest), and the emission mode is Super Pulse to reduce heat dispersion. It is applied to the mucosal surface without blood supply at the lower edge of the middle turbinate for 2 minutes on each side, totaling only 1.2 seconds of cumulative laser emission. Compared to the experimental group using 2W energy with continuous irradiation for 2 minutes, the total energy release difference in the sham surgery group is only 1/400 of the experimental group (2W120sec/0.5W1.2sec). This is to produce the sound, light, and tactile effects of the laser, but without sufficient energy transfer to cause high-temperature mucosal changes and tissue alterations, serving as a high-quality sham surgery control group.
  Arms: Sham surgery

SUMMARY:
This clinical trial aims to learn if laser posterior nasal nerve neurolysis can treat chronic rhinitis in adults. It will also learn about the safety of laser posterior nasal nerve neurolysis. The main questions it aims to answer are:

1. Does laser posterior nasal nerve neurolysis improve chronic rhinitis symptoms?
2. What side-effects or complications do participants have after laser posterior nasal nerve neurolysis?

Researchers will compare laser posterior nasal nerve neurolysis to a placebo(a sham surgery with the same device and sound to see if laser posterior nasal nerve neurolysis works to treat chronic rhinitis.

Participants will

1. Receive laser posterior nasal nerve neurolysis in the office as local anesthesia surgery.
2. Visit the clinic in the first week, first month, and 3rd months after the surgery.
3. Record their symptom scores before the surgery and during each follow-up visit.

DETAILED DESCRIPTION:
Chronic rhinitis is a highly prevalent condition characterized by symptoms such as nasal congestion, rhinorrhea, postnasal drip, nasal itching, and sneezing. First-line treatments typically include nasal irrigation, intranasal corticosteroids, intranasal anticholinergics, oral antihistamines, or topical decongestants. However, many patients fail to achieve satisfactory therapeutic outcomes through pharmacological interventions alone, resulting in significant impairment of quality of life and productivity.

In addition to pharmacotherapy, various surgical approaches have been proposed, including inferior turbinate reduction (partial or submucosal resection), radiofrequency inferior turbinate ablation (RFIT), microdebrider-assisted turbinoplasty, vidian neurectomy, and posterior nasal neurectomy or ablation. Vidian neurectomy is infrequently employed due to potential complications, including hemorrhage, malar and maxillary discomfort, and dry eye symptoms. While the introduction of endoscopic posterior nasal neurectomy has addressed some of these complications (malar and maxillary discomfort), patients may still experience dry eye.

In 2022 and 2023, the American Rhinologic Society (ARS) and the American Academy of Otolaryngology-Head and Neck Surgery (AAO-HNS) issued statements supporting the use of posterior nasal nerve neurolysis (PNNN) for the treatment of chronic rhinitis. These statements indicate that posterior nasal nerve neurolysis techniques, such as radiofrequency ablation and cryotherapy, have been utilized to disrupt the posterior nasal nerve in the sphenopalatine foramen region of the posterior middle meatus.

The application of CO2 laser for posterior nasal nerve cauterization has not yet been evaluated in large-scale randomized controlled clinical trials. In otolaryngological surgery, this laser is widely employed in pharyngolaryngeal procedures, vocal cord surgery, oral mucosal surgery, and intranasal and turbinate surgeries due to its excellent hemostatic properties and precision.

Therefore, the investigators propose this research protocol to conduct a randomized controlled clinical trial to determine whether posterior nasal nerve cauterization using CO2 laser can effectively control chronic rhinitis symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old
* Chronic rhinitis symptoms for at least 6 months that have not responded effectively to medication (should include at least Intranasal corticosteroid (ICS) combined with intermittent use of oral antihistamine and, as needed, combination nasal spray) or where medication has not provided sustained improvement
* Total rTNSS ≥ 5 with Moderate to severe rhinorrhea symptoms (24-hour reflective Total Nasal Symptom Score [rTNSS] rhinorrhea score of 2-3) and mild to severe nasal congestion symptoms (rTNSS nasal congestion score of 1-3)
* All enrolled patients routinely undergo endonasal endoscopic examination, or have had a sinus CT within the past month confirming no significant rhinosinusitis."

Exclusion Criteria:

* Obstructive anatomical abnormalities limiting access to posterior nasal passages
* Nasal anatomical changes due to previous sinus or nasal surgery or injury
* Ongoing nasal or sinus infection
* History of severe dry eye, chronic epistaxis, rhinitis medicamentosa, or head and neck radiotherapy
* Self-reported history of bleeding tendency
* Current use of anticoagulants with inability to discontinue
* Previous chronic rhinitis surgery
* History of poor wound healing after head, neck, or throat surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-06 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in chronic rhinitis score | From the date of randomization and every three months after intervention is performed on 3, 6, 9, and 12 months post intervention.
  The investigators will use reflective total nasal symptom score, (rTNSS, 0-12, the higher the worse) and Nasal Obstruction Symptom Evaluation(NOSE, 0-20, the higher the worse) to compare the chronic rhinitis symptoms before and after the intervention.

SECONDARY OUTCOMES:
Complications of the intervention | From the date of randomization and every three months after intervention is performed on 3, 6, 9, and 12 months post intervention.
  The investigators will document all the self-reported and observed complications after the intervention.

OTHER OUTCOMES:
Change in sleep quality and day time sleepiness scale | From the date of randomization and every three months after intervention is performed on 3, 6, 9, and 12 months post intervention.
  The investigators will compare the Pittsburgh Sleep Quality Index, (PSQI, 0-21, the higher the worse the sleep) and Epworth sleepiness Scale, (ESS, 0-24, with over 11 indicate sleepy, the higher the worse) of the enrolled patients before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lee JT, Abbas GM, Charous DD, Cuevas PDMM, Goktas PDMO, Loftus PA, Nachlas NE, Toskala EM, Watkins JP, Brehmer PDMD. Clinical and Quality of Life Outcomes Following Temperature-Controlled Radiofrequency Neurolysis of the Posterior Nasal Nerve (RhinAer) for Treatment of Chronic Rhinitis. Am J Rhinol Allergy. 2022 Nov;36(6):747-754. doi: 10.1177/19458924221109987. Epub 2022 Jul 11. PMID 35818709
- [Background] Takashima M, Stolovitzky JP, Ow RA, Silvers SL, Bikhazi NB, Johnson CD. Temperature-controlled radiofrequency neurolysis for treatment of chronic rhinitis: 12-month outcomes after treatment in a randomized controlled trial. Int Forum Allergy Rhinol. 2023 Feb;13(2):107-115. doi: 10.1002/alr.23047. Epub 2022 Jul 5. PMID 35714267
- See also: Position Statement: PNN Ablation for the Treatment of Chronic Rhinitis — https://www.entnet.org/resource/position-statement-posterior-nasal-nerve/